CLINICAL TRIAL: NCT05113862
Title: A Phase-I, Double-blind, Randomized, Vehicle-controlled, Dose-finding, Safety Study of a Synthetic Nanoparticle-based, T Cell Priming Peptide Vaccine Against SARS-CoV-2 in Healthy Adults in Switzerland
Brief Title: A Phase-I Study of a Nanoparticle-based Peptide Vaccine Against SARS-CoV-2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gylden Pharma Ltd (Industry)
Collaborators: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other); University of Lausanne Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: naNO-COVID
Record Dates: First submitted 2021-11-05; First posted 2021-11-09 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2022-11

CONDITIONS: Coronavirus; SARS-CoV-2 Infection; COVID-19
Keywords: Coronavirus; SARS-CoV-2; COVID-19; T-cell priming; COVID vaccine; nanoparticle; T-cell vaccine
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: * This trial is double-blinded (blinded to investigators and participants)
  * Blinding will be maintained for the duration of the study
  * All allocations will remain coded to all volunteers and investigators. An independent pharmacy team at CHUV will label the vaccine and comparator doses with coded participant numbers but will not have access to the identifier list linking the code to the participant identity. All vaccine and comparator doses will be prepared and labelled away from investigators and stored in identical conditions.
  * The appearance of the comparators and doses will be identical. The solutions of both are indistinguishable within the dosage group and thus no shielding of the solution colour is needed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LD Vehicle GNP (Sham Comparator): Low dose (LD) comparator (2.5nmol) - gold nanoparticle (12.8ug) without peptides
  Interventions: Biological: LD Vehicle-GNP
- LD PepGNP-Covid19 (Experimental): Low dose (LD) peptide vaccine (2.5nmol) - gold nanoparticle (12.8ug) plus peptides
  Interventions: Biological: LD PepGNP-Covid19
- HD Vehicle GNP (Sham Comparator): High dose (HD) comparator (7.5nmol) - gold nanoparticle (38.3ug) without peptides
  Interventions: Biological: HD Vehicle-GNP
- HD PepGNP-Covid19 (Experimental): High Dose (HD) peptide vaccine (7.5nmol) - gold nanoparticle (38.3ug) plus peptides
  Interventions: Biological: HD PepGNP-Covid19

INTERVENTIONS:
Biological: LD Vehicle-GNP — Two intradermal injections in the upper arm spaced 21 days apart
  Arms: LD Vehicle GNP
Biological: LD PepGNP-Covid19 — Two intradermal injections in the upper arm spaced 21 days apart
  Arms: LD PepGNP-Covid19
Biological: HD Vehicle-GNP — Two intradermal injections in the upper arm spaced 21 days apart
  Arms: HD Vehicle GNP
Biological: HD PepGNP-Covid19 — Two intradermal injections in the upper arm spaced 21 days apart
  Arms: HD PepGNP-Covid19

SUMMARY:
This trial is Stage 2 of a 2-part adaptive trial. The study aims to investigate the safety of 2 doses of a T-cell priming specific cocktail of Coronaviruses peptides mounted on a gold nanoparticle.

Note: Stage 1 of the 2-part adaptive trial, testing a specifically selected mix of Dengue virus peptides, commenced Aug 2021. This is now in follow up (NCT04935801).

DETAILED DESCRIPTION:
Despite drastic quarantine measures, SARS-CoV-2 continues to propagate and threaten global economies and healthcare systems. There is universal consensus on the need for vaccination to protect against complications, reduce viral shedding and therefore prevent severe manifestation of disease and reduce hospitalisations.

Coronavirus harbours the potential to become a seasonal disease. It is moving towards being a ''new flu'' with potential perennial circulation and continuously evolving Variants of Concern (VOCs), needing diverse vaccines to control it. The Global Vaccine Alliance, GAVI, has specifically advocated for vaccine diversity as a means to ensure equality and access as well as a means of maximising scalability.

Nanoparticle antigen delivery systems have been developed to enrich specific targeting of immune receptors. These carrier systems are designed to facilitate antigen uptake and processing by antigen presenting cells (APCs), as well as to control antigen release and protect them from premature proteolytic degradation. This more targeted response also allows to reduce the effective antigen dose (to nanomoles) and mimic a replicating infection with zero risk of developing the infectious disease.

The hypotheses are listed below:

1. The scale of the COVID-19 pandemic requires multiple vaccine candidates to ensure democratic and rapid access to protection by:

   * Providing a range of vaccine choices tailored to variations in immunological profiles across demographics as well as suited to environments with various levels of resources (cold chain etc).
   * Distributing and parallelizing manufacture, to speed up scale, avoid reagent stock limitations and dilute monopolies.
2. The ability for SARS-CoV-2 to mutate, requires multiple vaccine candidates to ensure robust and sustainable protection. Vaccines with a range of epitopes and immune targets provide immunological diversity and reduce vulnerability to mutant escape.
3. Nanotechnology fulfils the needs of a COVID vaccine by being a rapidly scalable and modular platform.
4. Humoral immunity may be transient and insufficient against emerging variants of SARS-CoV-2.
5. Cellular immunity against SARS-CoV-2 is lasting and associated with recovery in COVID-19.

The proposed vaccine of this trial specifically seeks to diversify the immunological target response by carefully curating an MHC-I binding antigen cocktail from the SARS viruses ligandome and loading it onto a robust nanoparticle for controlled release and coupled T-cell immunostimulation. It also specifically seeks to avoid generating a humoral response, which has the potential to be transient and even detrimental in certain cases.

For this second stage of the trial, the objectives are are follows:

Primary:

To evaluate the safety and reactogenicity of two intradermal injections of two different doses of the investigational COVID peptide T-cell inducing vaccine (PepGNP-Covid19) administered to healthy volunteers in Switzerland as a:

1. candidate vaccine for the prevention of COVID-19
2. proof-of-concept for a rapidly scalable modular peptide vaccine platform.

Secondary:

1. To assess the evidence of a CD8 T-cell mediated immune response as a surrogate of protection against severe COVID-19 disease using a novel peptide set-point vaccine in healthy adults.
2. To assess the presence of an antibody mediated response.

For naNO-COVID, a total of 26 eligible participants will be randomised into the following groups:

Group 1 (n=13) 10 low dose (LD) PepGNP-Covid19 (2.5nmol peptide +12.8ug) + 3 Comparator.

Group 2 (n=13) 10 high dose (HD) PepGNP-Covid19 (7.5nmol + 38.3ug) + 3 Comparator.

Thus, 20/26 vaccine and 6/26 Comparator controls. Allocations of vaccine vs bpC for each group are double-blinded. Each arm will be staggered into a ''Pioneer'' group (3/13 participants) followed a week later after a safety review by the remaining 10/13 ''Followers''.

This is the second stage of a 2-stage study investigating the safety of 2 vaccines from a T-cell priming vaccine platform for emerging diseases. (stage 1 = naNO-Dengue, stage 2 = naNO-COVID).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 45 years on the day of inclusion
* Participant signed informed consent
* Residing in Switzerland

Exclusion Criteria:

* Participant is pregnant, lactating or of childbearing potential
* Participation in the 4 weeks preceding the first trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device or medical procedure.
* Receipt of any vaccine (including vaccine against COVID) in the 4 weeks preceding the first trial vaccination (excluding influenza vaccination which may be received 2 weeks prior to the first vaccination), or planned receipt of any vaccine in the 4 weeks following each trial vaccination.
* Positive SARS-CoV2 test in the 4 weeks preceding the first trial vaccination.
* Receipt of immunoglobins, blood or blood-derived products in the past 3 months.
* Known, or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy.
* Self-reported or documented seropositivity for human immunodeficiency virus (HIV), hepatitis B natural infection, (HBcAb positive serology) or hepatitis C.
* Known systemic hypersensitivity to any of the vaccine components (e.g gold,) or history of a life-threatening reaction to vaccines.
* Current alcohol abuse or drug addiction (reported or suspected)
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion.
* Thrombocytopenia or any coagulation disorder
* Identified as an Investigator or employee of the Investigator or study centre with direct involvement in the proposed study, or identified as an immediate family member (i.e parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study (i.e in the employment of the Tropivac Clinic or DFRI unit at Unisante).
* Refusal to be informed in the event that relevant results concerning the participant's health are revealed.

The following events constitute contraindications to the administration of the investigational product on the day of planned vaccination: The participant must be followed until resolution of the event as with any medical event and may be considered for vaccination at a later date (maximum 14 days later) or withdrawn at the discretion of the Investigator. Delays due to these events do not constitute a protocol deviation.

* Temperature of >37.5°C at the time of vaccination
* Acute disease at the time of vaccination (defined as the presence of a moderate or severe illness with or without fever according to investigator's judgment. All vaccines can be administered to persons with a minor illness such as diarrhoea, mild upper respiratory infection with or without low-grade febrile illness, i.e. axillary temperature of ≤ 37.5°C).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Safety: Solicited local & systemic AEs | Through 14 days after prime or boost vaccination
  Number of volunteers overall and in each dose group with local or systemic vaccine reactogenicity, based on evaluation of solicited adverse events (AEs) recorded on subject memory aids or during clinical assessments
Safety: Unsolicited AEs | Study Days 0-180 or through termination visit, if terminated early
  Number of volunteers overall and in each dose group with unsolicited vaccine-associated adverse events (AEs) in each dose group
Safety: SAEs | Study Days 0-180 or through termination visit, if terminated early
  Number of volunteers overall and in each dose group with vaccine-associated serious adverse events (SAEs)
Safety: Adverse Events of Special Interest (AESI) | Study Days 0-180 or through termination visit, if terminated early
  Number of volunteers overall and in each dose group with vaccine-associated adverse events of special interest (AESIs)

SECONDARY OUTCOMES:
Immunogenicity: Proportion of participants with CD8-T cell specific to PepGNP-Covid19 | Study Days 0-180 or through termination visit, if terminated early
  Frequency of CD8+ T cells specific for individual CTL peptides by flow cytometry, using ex vivo MHC I dextramer staining and activation-induced markers (AIM)
Proportion of participants becoming seropositive (antibodies against SARS-CoV-2) | Study Days 0-180 or through termination visit, if terminated early
  Geometric mean titre and geometric mean fold rise of antibodies against SARS-CoV2 as determined by Enzyme-linked Immunosorbent Assay (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Blaise Genton, Prof., Principal Investigator — Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland
Locations (1):
- Center for Primary Care and Public Health (Unisante), Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The Investigators will be involved in writing and /or reviewing drafts of the manuscripts, abstracts, press releases and any other publications arising from the study.
  Apart from the obvious flaws to conduct of the study, which may preclude data publication, safety and efficacy data will be published under the supervision and authorisation of the PI and Sponsor.
  Publication will include as much individual level data as possible to ensure reproducibility of results without compromising participant privacy.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 12 months of study completion
Access Criteria: Peer-reviewed publication

REFERENCES:
- [Derived] Besson J, Audran R, Karlen M, Miauton A, Hajjami HM, Warpelin-Decrausaz L, Sene L, Schaufelberger S, Faivre V, Faouzi M, Hartley MA, Spertini F, Genton B. A gold nanoparticle/peptide vaccine designed to induce SARS-CoV-2-specific CD8 T cells: a double-blind, randomized, phase 1 study in Switzerland. BMC Infect Dis. 2025 Apr 7;25(1):472. doi: 10.1186/s12879-025-10844-3. PMID 40197245